CLINICAL TRIAL: NCT04348877
Title: Plasma Rich Antibodies From Recovered Patients From COVID19
Acronym: PRA-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hossam Fahmy, Professor of Faculty of Medicine, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P15/ 2020
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Disease (COVID-19)
Keywords: Egypt
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Antibody-Rich Plasma from COVID-19 recovered patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antibody-Rich Plasma (Other): 400 millimeter of Antibody-Rich Plasma from COVID-19 recovered patients will be transfused to patients with severe or immediately life-threatening COVID-19
  Interventions: Other: Antibody-Rich Plasma from COVID-19 recovered patients

INTERVENTIONS:
Other: Antibody-Rich Plasma from COVID-19 recovered patients — 400 millimeter of Antibody-Rich Plasma from COVID-19 recovered patients will be transfused to patients with severe or immediately life-threatening COVID-19

SUMMARY:
Prospective interventional study, single arm of purified convalescent plasma transfusion as an add on therapy for the standard of care treatment (national guideline) (Oseltamivir (75mg/12 hours for 5-10 days) and hydroxychroquine (400mg twice in first day, 200 twice for 4-9 days) ± Azithromycin 500mg daily for 5 days

DETAILED DESCRIPTION:
1. Selection of donor according to the eligibility criteria

   * Full medical history, concurrent medications, demographic data will be obtained.
   * Complete clinical assessment with special emphasis on assessment of resolution of symptoms
   * Body weight, height.
   * A confirmatory diagnostic test result (e.g., nasopharyngeal swab) at the time of illness or serological test for SARS-CoV-2 antibodies after recovery will be collected
   * COVID -19 PCR test by nasopharyngeal swab.
   * Complete blood count with differential counts
   * Viral screening (HBV, HCV, HIV & Syphilis): Conventional testing by chemiluminescence followed by nucleic acid testing (NAT)
   * Donor's written consent
2. Plasma collection:

   * Donor to be connected to microprocessor controlled plasmapheresis machine containing single use disposable kit for every donor.
   * A certain amount of blood is withdrawn by pump from the patient and immediately anticoagulated then centrifuged in the machine.
   * Blood components are separated into different layers according to the density of each component.
   * The plasma layer is collected and diverted into the collection bag while all other components are infused back to the patient, thus ending the first cycle.
   * Cycles are repeated until collecting a total of 400 ml of filtered plasma in the collection bag; that is one complete therapeutic dose for one patient in need.
3. Pathogen reduction/Viral inactivation by the Solvent/Detergent (S/D) method:

   * SD method is the gold standard for inactivation of enveloped viruses HBV, HCV and HIV. All these viruses have a lipid outer coat enveloping the nucleic acid.
   * Tri-N Butyl Phosphate (TNBP) acts as an organic solvent to remove lipids from the membranes of pathogens.Tween-20 is a non-ionic detergent that stabilizes TNBP and disrupts lipid bilayers, thus easing the extraction of lipids. Since the solvent is toxic, it is removed using a sterile vegetable oil (Castor oil).
4. Measuring remnants of TNBP:

   * By chromatography in Ain Shams Toxicology Center.
   * Concentration should be less than 10 ppm.
5. Screening phase for patients selection:

   • Obtaining informed consent: Written signed and dated informed consent will be obtained from each patient before being entered into the study. The investigator, or a person designated by the investigator, should fully inform the subject or, if the subject is unable to provide informed consent, the subject's legally acceptable representative, of all pertinent aspects of the trial. This will be obtained from each subject in accordance with the recommendation of the revised Declaration of Helsinki. The investigator will explain the nature, purpose and risks of the study. It will be clearly stated that the patient is free to withdraw from the study at any time for any reason without prejudice to future care, and with no obligation to give the reason for withdrawal.

   In case the patient is unable to provide his/her consent the legal guardian will give verbal approval on behaves of the patient and after he he/she will be well informed by the study design, procedure, risk and benefits over phone call.

   If it is difficult to reach the legal guardian, emergency approval will be obtained by Professional Legal Representative who will be the head authorities of the isolation hospital.
   * Full medical history, concurrent medications, demographic data will be obtained.
   * A thorough physical examination will be performed.
   * Body weight, height, BMI, vital signs (blood pressure, heart rate and temperature) and Blood oxygen saturation) will be recorded.
   * Chest x-ray and CT scan for chest will be recorded
   * Ventilation parameters to be recorded if ventilated
   * Laboratory to perform the following tests:

   Complete blood count with differential counts, Renal function tests (RFTs) (serum creatinine), Liver function tests (LFTs) (alanine amino transferase (ALT), aspartate amino transferase (AST), total and direct bilirubin), Coagulation test; prothrombin time and INR and D.dimer, HIV Ab, HCV Ab and HBV surface antigen (HBsAg), COVID -19 PCR test by nasopharyngeal swab. Urine pregnancy test for females.
6. Treatment phase for eligible patients:

   * Eligibility confirmed
   * Treatment with collected plasma in a dose of 400 ml on single therapeutic dose on Day1 as an add on therapy for the standard of care treatment (national guideline) (Oseltamivir (150mg/12 hours for 5-10 days) and hydroxychroquine (400mg twice in first day, 200 twice for 4-9 days) ± Azithromycin 500mg daily for 5 days.
   * The patient's health status, and the presence of adverse events will be assessed daily
   * Complete physical examination will be performed daily.
   * Vital signs (blood pressure, heart rate and temperature) will be recorded.
   * Follow-up CXR will be performed on daily and /CT scan will be performed as clinically indicated
   * Coagulation test; prothrombin time and INR and D.dimer will be re-reassessed on day 3, 7, and 14
   * HIV Ab, HCV Ab and HBV surface antigen (HBsAg) will be repeated at day 14
   * COVID -19 PCR test by nasopharyngeal swab will be repeated every 72 hours.
   * Post treatment period up to 30 days after end of treatment:

     * Vital signs (blood pressure, heart rate and temperature) will be recorded.
     * Symptoms and signs assessment will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 -80 years old
2. Must have laboratory confirmed COVID-19
3. Must have severe or immediately life-threatening COVID-19, Severe disease is defined as: Dyspnea,Respiratory frequency ≥ 30/min,Blood oxygen saturation ≤ 93%,Partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or lung infiltrates > 50% within 24 to 48 hours Life-threatening disease is defined as: respiratory failure, septic shock, and/or multiple organ dysfunction or failure
4. Must provide informed consent by patient or his/her legal guardian or Professional Legal Representative

Exclusion Criteria:

* Patient with mild or moderate COVID-19
* Participation in any investigational clinical study, other than observational, within the past 30 days; or plans to participate in such a study at any time from the day of enrollment until 30 days post-treatment in the current study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
viral COVID-19 clearance | 14 days
  Two successive negative COVID-19 PCR analysis tests 72 hours apart

SECONDARY OUTCOMES:
Decrease of radiological abnormalities | 14 days
  The percentage of decrease of radiological abnormalities at day 14
Clinical improvement | 14 days
  Clinical improvement in form of normal body temperature for 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No